CLINICAL TRIAL: NCT05982834
Title: Disitamab Vedotin Combined With Fruquintinib and Tislelizumab in Second-line Treatment for HER2-positive Metastatic Gastric Cancer: A Prospective Phase Ib/II Study
Brief Title: Disitamab Vedotin, Fruquintinib and Tislelizumab in Second-line Treatment for HER2-positive MGC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, Principal Investigator, Clinical Professor of the Department of Medical gastrointestinal oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-RCPF
Record Dates: First submitted 2023-05-19; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Gastric Cancer; Immunotherapy
MeSH Terms: interventions — HMPL-013; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin combined with fruquintinib and Tislelizumab (Experimental)
  Interventions: Drug: Disitamab Vedotin combined with fruquintinib and Tislelizumab

INTERVENTIONS:
Drug: Disitamab Vedotin combined with fruquintinib and Tislelizumab — Disitamab Vedotin 2.5mg/m2 ivgtt d1,15, fruquintinib 4mg qd po d1-21 and Tislelizumab 300mg ivgtt,q4w

SUMMARY:
At present, there is no anti-HER2 therapy recommended by guidelines for second-line treatment of advanced gastric cancer with HER2-positive or HER2-overexpression, and combined with anti-angiogenic drugs are mainly used. Disitamab Vedotin is an anti-HER2 ADC, and its cytotoxic drugs are also anti-microtubule formation as the main mechanism of drugs. Fruquintinib is an anti-vascular TKI drug. In addition, according to the results of KEYNOTE-811, patients with HER2-positive advanced gastric cancer benefit significantly from immunotherapy, so the investigators hope to explore the possibility of immunotherapy in second-line treatment of HER2-positive advanced gastric cancer. Therefore, the study plans to enroll HER2-positive patients who have failed first-line therapy and explore the efficacy of the regimen of Disitamab Vedotin combined with fruquintinib combined with Tislezumab in second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. older than18 years of age, gender not limited;
2. the histologic diagnosis of the stomach or gastroesophageal junction adenocarcinoma;
3. immunohistochemical HER2 2 + 3 + or HER2, FISH is positive;
4. at least have a measurable lesions (10 mm or higher spiral CT scan, RECIST 1.1 standard);
5. First-line treatment failure of fluorouracil and the platinum, or to accept containing fluorouracil and platinum adjuvant chemotherapy in patients with recurrence after 6 months;
6. ECOG 0-2, expected survival for 3 months or more;
7. the subjects treated with other damage has been restored, accepting radiotherapy should be ended more than 3 weeks;
8. major organs function is normal, the group within 1 week before the lab test results meet the following criteria: (1) The standard of blood routine examination shall meet:

   1. HB≥80g/L;
   2. ANC ≥1.5×109/L;
   3. PLT ≥75×109/L (2) Biochemical examination shall meet the following standards:

   a. Total bilirubin BIL < 1.25 * upper limit of normal (ULN) B. the ALT and AST acuities were 2.5 * ULN. C. serum creatinine (Cr) of 1.5 or less * ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft - Gault formula)
9. participants voluntarily participate in this study, and signed by himself or agent informed consent; Patient compliance is good, can cooperate with the relevant examination, treatment and follow-up.

Exclusion Criteria:

1. history of other malignant tumors within 3 years, have cured except cervical carcinoma in situ or skin basal cell carcinoma;
2. with brain or meningeal metastasis;
3. associated with gastrointestinal obstruction, gastrointestinal bleeding (defecate occult blood + + + and above) or perforation;
4. with active, or have a history and possible recurrence of autoimmune disease of the subjects (such as: Systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or those at high risk (such as those who have received an organ transplant requiring immunosuppressive therapy), However, patients with vitiligo, psoriasis, alopecia, or Grave's disease who did not require systemic treatment within the last 2 years, or patients with hypothyroidism who only needed thyroid hormone replacement therapy, and patients with type I diabetes who only needed insulin replacement therapy could be enrolled;
5. now with interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung diseases, radiation pneumonia;
6. within 4 weeks before delivery for the first time to participate in any other drug clinical research (the use of test drugs shall prevail), unless the participant observation (non intrusive) clinical research;
7. within 4 weeks before the first dose of study treatment used immunosuppressive drugs, Does not include nasal, inhalation or other routes of topical corticosteroids or physiological doses of systemic corticosteroids (i.e., not exceeding 10 mg/ day of prednisone or equivalent doses of other corticosteroids), or short-term (not exceeding 7 days) use of corticosteroids for the prevention or treatment of non-autoimmune allergic diseases;
8. within 4 weeks before the first dose of study treatment or accept the live attenuated plan during the study period. Note: Inactivated virus vaccines for injectable seasonal influenza are permitted for up to 4 weeks prior to initial administration; But live attenuated influenza vaccines are not allowed;
9. within 4 weeks before the first dose of study treatment received major surgery, open chest or craniotomy laparotomy or expected during the research and treatment need to accept of this study major surgery.
10. infected with human immunodeficiency virus (HIV) disease (i.e., an HIV positive), or with other acquired, congenital immunodeficiency disease, or has a history of history of organ transplantation, or stem cell transplantation;
11. chronic active hepatitis b or active active hepatitis c, hepatitis b virus carriers, stable after drug treatment of hepatitis b (DNA drop degree is not higher than 200 iu/mL or copy number Copies <1000copies/mL) and cured hepatitis C patients (HCV RNA test negative) could be included;
12. with known active tuberculosis;
13. first before 4 weeks with severe infections, or 2 weeks before appear active infection need oral or intravenous antibiotic therapy patients;
14. symptomatic congestive heart failure (New York heart association grade II - IV) or symptomatic or poorly controlled arrhythmia.
15. even give specification treatment still uncontrolled arterial blood pressure (systolic blood pressure or greater acuity 160 MMHG or diastolic blood pressure, 100 MMHG).
16. within 6 months before the selected treatment occurred any arterial thromboembolic events, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.
17. within 3 months before the group with deep vein thrombosis, pulmonary embolism, or any other serious history of thromboembolism (implantable venous infusion port source sex or catheter thrombosis, or superficial venous thrombosis were not regarded as a "severe" thromboembolism).
18. always have a clear history of neurological or psychiatric disorders, such as memory, epilepsy, dementia, compliance, or the peripheral nervous system disorder;
19. alcohol dependence or nearly 1 year has a history of drug or drug abuse;
20. pregnancy or lactation women; Those who are fertile but do not take adequate contraceptive measures;
21. may lead to the following results of other acute or chronic diseases, mental illness or abnormal laboratory values: participated in or study drug dosage associated with an increased risk, or interfere with the interpretation of results, and according to the researcher's judgment will be patient as does not conform to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 8 weeks, up to 1 year.
  the proportion of patients whose tumor dcrease to a certain size and remained for a certain period of time, including those with complete response(CR) and partial response (PR).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No